CLINICAL TRIAL: NCT07229105
Title: Comparative Effectiveness of Remineralization Agents on Attachment-Associated Demineralization in Clear Aligner Patients: A 6-Month DIAGNOdent-Based Observational Study
Brief Title: Comparative Effectiveness of Remineralization Agents on Attachment-Associated Demineralization in Clear Aligner Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Banu Kılıç, Assistant Professor, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 09/15
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: White Spot Lesions; Demineralization; Dental Caries; Orthodontic Treatment
Keywords: clear aligners; Orthodontic Attachments; DIAGNOdent; White Spot Lesions; White Spot Lesion
MeSH Terms: conditions — Dental Caries | interventions — Bifluorid 12

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Control (No Intervention): The participants used standard fluoride toothpaste (1450 ppm) twice daily, with no additional remineralization protocol.
- Group B: Casein Phosphopeptide-Amorphous Calcium Phosphate (Experimental): In addition to standard fluoride toothpaste, participants applied GC Tooth Mousse (CPP-ACP) to their clear aligners once daily for 15 minutes before bedtime.
  Interventions: Device: GC Tooth Mousse
- Group C: Nano-Hydroxyapatite (Experimental): Professional in-office application of 5% nHAp gel at baseline, 1, and 3 months, combined with daily home application of 1% nHAp gel into aligners.
  Interventions: Device: Nano-Hydroxyapatite Gel
- Group D: Professional Fluoride Varnish (Experimental): Professional application of 5% sodium fluoride varnish (ProShield) applied to attachment margins at baseline and 3 months.
  Interventions: Drug: Sodium Fluoride varnish

INTERVENTIONS:
Device: GC Tooth Mousse — Participants applied a pea-sized amount of GC Tooth Mousse into each aligner once daily before bedtime. They wore the aligners with the mousse for 15 minutes and were instructed not to rinse for 30 minutes post-application.
  Other Names: CPP-ACP Paste
  Arms: Group B: Casein Phosphopeptide-Amorphous Calcium Phosphate
Device: Nano-Hydroxyapatite Gel — A combined protocol involving: 1) Professional in-office application of 5% nHAp gel (BioWhiten ProOffice) at baseline, 1 month, and 3 months; and 2) Daily home application of 1% nHAp gel (Biowhiten Nanocare) into aligners every night before sleep.
  Other Names: BioWhiten ProOffice and Nanocare
  Arms: Group C: Nano-Hydroxyapatite
Drug: Sodium Fluoride varnish — Professional application of 5% sodium fluoride varnish (ProShield) to all tooth surfaces, with special attention to attachment margins, at baseline and 3 months. The varnish was left for 1 minute contact time before removal, with instructions not to eat/drink for 2 hours.
  Other Names: ProShield Varnish
  Arms: Group D: Professional Fluoride Varnish

SUMMARY:
Background/ Objectives: Clear aligner attachments increase the risk of white spot lesions (WSL), with a 35.5% incidence in adolescents. The number of anterior attachments is an independent risk factor (OR=2.192). Despite 17 million patients treated worldwide, no study has quantitatively assessed demineralization around attachment margins. To compare the effectiveness of CPP-ACP, nano-hydroxyapatite (nHAp), and fluoride varnish versus a control for attachment-associated demineralization using DIAGNOdent monitoring.

Methods: This prospective observational study evaluated 52 patients; 45 were enrolled, and 40 completed after five pre-baseline withdrawals. Participants were allocated to four groups (n=10 each): Group A (control, fluoride toothpaste), Group B (CPP-ACP daily), Group C (nHAp professional + home gel), and Group D (fluoride varnish quarterly). DIAGNOdent measurements were taken around attachments at baseline, 1, 3, and 6 months. Linear mixed-effects models analyzed group differences (p<0.05).

DETAILED DESCRIPTION:
DIAGNOdent Measurement Protocol Calibration and Standardization The DIAGNOdent pen (KaVo, Biberach, Germany) was calibrated before each measurement session according to the manufacturer's instructions using a ceramic standard[18]. A single calibrated examiner performed all measurements to ensure consistency. Intra-examiner reliability was assessed using intraclass correlation coefficient (ICC) with two-way mixed model, absolute agreement, calculated from 30 repeated measurements at 10 randomly selected attachment sites (ICC = 0.85, 95% CI: 0.79-0.91).

Measurement Technique A standardized measurement protocol was employed for all DIAGNOdent assessments. Teeth were air-dried for 5 seconds prior to measurement, and the probe tip was positioned perpendicular to the enamel surface to ensure consistent readings. Four measurements were obtained per attachment site at the mesial, distal, gingival, and occlusal margins. Three measurement passes were performed at each site, with the maximum value recorded to represent the most advanced demineralization present. Measurements were conducted at four timepoints: baseline (T0), 1 month (T1), 3 months (T2), and 6 months (T3).

ELIGIBILITY:
Inclusion Criteria:

* Age 16-45 years
* Active clear aligner treatment with minimum 6 months remaining
* Presence of ≥10 attachments on anterior teeth and premolars
* Good general health
* Commitment to prescribed aligner wear (20-22 hours/day)

Exclusion Criteria:

* Active carious lesions
* Periodontal disease
* Fluorosis or enamel hypoplasia
* Current fluoride supplement use beyond standard toothpaste
* Pregnancy or lactation
* Systemic conditions affecting salivary flow

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Change in Enamel Demineralization (DIAGNOdent values). | Baseline (T0) to 6 months (T3).
  Measurements taken using DIAGNOdent pen around attachment margins. Validated cut-off values: 0-12 sound, 13-24 initial, >25 advanced.

SECONDARY OUTCOMES:
Temporal Changes in Enamel Mineralization | 1 month (T1) and 3 months (T2)
  Evaluation of DIAGNOdent values at intermediate time points to assess the progression or regression patterns (e.g., continuous improvement vs. biphasic response) of demineralization.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and analysed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication
Access Criteria: Researchers can contact the corresponding author.